CLINICAL TRIAL: NCT03747445
Title: Microstructural Analysis of Ingestive Behavior After Roux-en-Y Gastric Bypass - a Prospective Controlled Exploratory Pilot Study Using a Novel Drinkometer to Measure Liquid Lunch Intake
Brief Title: Microstructural Analysis of Ingestive Behavior After Roux-en-Y Gastric Bypass - Pilot
Status: Completed | Type: Observational
Sponsor: Marco Bueter (Other)
Collaborators: Department of Psychology and Program in Neuroscience, Florida State University, Tallahassee, FL, USA (Unknown)
Responsible Party: Sponsor-Investigator, Marco Bueter, Assistant Professor, PhD, Head of Bariatric Program, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2017-00756-2
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Meal; Obesity, Morbid; Food Deprivation; Bariatric Surgery; Roux-en-y Gastric Bypass; Ingestive Microstructure; Drinking Behavior; Drinkometer
MeSH Terms: conditions — Obesity, Morbid; Drinking Behavior | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Roux-en-Y gastric bypass patients: severely obese non-diabetic adult female patients scheduled for RYGB
  Interventions: Procedure: Roux-en-Y gastric bypass
- Normal weight controls: normal weight healthy non-diabetic adult females
- Obese controls: Severely obese non-diabetic adult female patients not scheduled for RYGB

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — laparoscopic surgical procedure
  Groups: Roux-en-Y gastric bypass patients

SUMMARY:
The ability to assess ingestion in fine detail over the time course of a liquid meal allows for comparison of early and late meal features of drinking and may help dissociate manipulations (surgical, neural, pharmacological, etc.) that affect orosensory properties from those that are modulating postoral processes in the control of intake.

The aim of the study is to asses microstructural changes in liquid meal intake over 1-year in severely obese patients after Roux-en-Y gastric bypass (RYGB).

DETAILED DESCRIPTION:
Introduction

Bariatric surgery (BS) is currently the most effective treatment of severe obesity. BS has a pleiotropic effect on the body, involving changes in basic metabolic rate, gut hormone and bile acid levels, intestinal nerve signaling and microbiota composition. Overall, patients report to eat less, to feel less hungry and they often change their taste preferences. Initial insights on food intake and appetite can be provided by indirect measures such as verbal report of energy intake, food diaries, and dietary recall questionnaires. However, indirect measures are vulnerable to inaccuracy and, at best, only offer an estimate of the target behavior. Such methodological limitations can be improved by complementing existing findings with direct measures of feeding and drinking. There are only very few studies to date that have applied direct measures of ingestive behavior in BS patients. These studies focused mainly on macronutrient composition within a cafeteria diet and on some motivational aspects of appetite behavior. This might be due to the fact that the assessment of the temporal organization of ingestive behavior within a meal in humans poses significant methodological and conceptual challenges to researchers and study design. The investigators have recently developed and validated a novel drinkometer for humans, which may have great utility in investigations of the specific behavioral variables that underlie the dysregulation of appetite control in morbid obesity, and also to specify neural effects of various medical or surgical weight-loss interventions.

The aim of this exploratory pilot study is to observe the ingestive microstructure of a liquid meal intake before and several occasions after RYGB. Observed values may serve as basis for designing future observational studies in the field of obesity research.

Methods

Prospective observational controlled cohort pilot study in severely obese patients scheduled for RYGB. 11 patients and 10 normal-weight controls will be recruited to consume a calorically dense standardized refrigerated liquid meal (product: Resource 2.0+fibre, Nestle, Vevey, Switzerland) in a food deprived state, until reaching satiety. The novel drinkometer will be used to measure ingestive microstructure and overall intake, and anthropometric parameters (weight, height) will be measured as well. Visual analogue scales will be used to assess self-reported hunger, thirst, fullness, taste preference and participants will estimate their intake at the end of each session. Time points for patients: pre-operatively, postoperative 1 week, 1-3-6-12 months. Time points for control group: baseline, 1-3-12 months. Due to major differences in ingestive microstructure, only female participants will be included in the study.

Satistical analysis

The drinkometer data will be processed and filtered by an in-house developed algorithm in Matlab 2017 software. Results will be analysed using descriptive statistics, as well as ANOVA, t-tests and Wilcoxon signed rank test in R software version 3.5.1.

Potential outcomes

Any comprehensive understanding of how BS affects food intake requires a detailed analysis of the ingestive behavior itself, not simply the measurement of the outcome of the behavior. In other words, the information on how the food is consumed is equally or even more important than the information on how much food has been ingested. To the best of our knowledge, this is the first time that drinking microstructure in humans will be recorded and analyzed after BS. Results will inform on the range of values that can be observed in this patient population and will serve as a basis to accurately power future studies in this field. Further, this exploratory study may generate hypothesis on behavioral changes that occur following BS. Any treatment that affects total intake - e.g. BS - can be entirely viewed as function of its single components such as size and number of sucking bursts which then can provide relevant information e.g. on the motivational aspects of the ingestive behavior. The investigators expect to find no difference in the ingestive behavior between patients before and after RYGB and in comparison to lean controls when the high-sugar high-fat stimulus is consumed for the first time. The investigators also do not expect an effect of RYGB on the number of sucking events within the first minute of the test session. As initial suck rate reflects the consummatory behavior in response to a given stimulus and thus indicate the initial motivational state toward this stimulus, the lack of RYGB-induced changes in this microstructural parameter would suggest that RYGB does not change the palatability of the stimulus. In line with this, the investigators further expect that suck rate during consumption of the fluid will decrease as a function of meal progress and with progressing postoperative time in patients after RYGB, but not in lean controls. Regardless of which outcomes are obtained, this innovative experiment will be a critical and a novel test of the explicit experience of humans with a high-sugar high-fat liquid meal after RYGB and its potential role for the understanding possible mechanisms determining postoperative outcomes, such as weight loss.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide inform consent
* treatment group: scheduled for RYGB for severe obesity
* control group: normal weight, healthy general condition

Exclusion Criteria:

* lactose intolerance
* diabetes
* immunosuppression
* pregnancy / lactation
* use of weight-loss medication

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult females with severe obesity and scheduled to undergo RYGB
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
change in microstructure of ingestive behavior of 1 liquid meal | baseline, 1 week, 1-3-6-12 months
  recording of meal intake by the drinkometer

SECONDARY OUTCOMES:
change in self-reported hunger, thirst, fullness, taste preference, estimated consumption | baseline, 1 week, 1-3-6-12 months
  visual analogue scale (0-100 mm, higher number refer to stronger feeling/higher liking)
body mass index | baseline, 1 week, 1-3-6-12 months
  weight/height measurements

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bueter, MD, PhD, Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gero D, File B, Justiz J, Steinert RE, Frick L, Spector AC, Bueter M. Drinking microstructure in humans: A proof of concept study of a novel drinkometer in healthy adults. Appetite. 2019 Feb 1;133:47-60. doi: 10.1016/j.appet.2018.08.012. Epub 2018 Sep 1. PMID 30179650
- [Background] Gero D, Steinert RE, le Roux CW, Bueter M. Do Food Preferences Change After Bariatric Surgery? Curr Atheroscler Rep. 2017 Sep;19(9):38. doi: 10.1007/s11883-017-0674-x. PMID 28779431
- [Background] Mathes CM, Bohnenkamp RA, Blonde GD, Letourneau C, Corteville C, Bueter M, Lutz TA, le Roux CW, Spector AC. Gastric bypass in rats does not decrease appetitive behavior towards sweet or fatty fluids despite blunting preferential intake of sugar and fat. Physiol Behav. 2015 Apr 1;142:179-88. doi: 10.1016/j.physbeh.2015.02.004. Epub 2015 Feb 3. PMID 25660341
- [Background] Spector AC, Klumpp PA, Kaplan JM. Analytical issues in the evaluation of food deprivation and sucrose concentration effects on the microstructure of licking behavior in the rat. Behav Neurosci. 1998 Jun;112(3):678-94. doi: 10.1037//0735-7044.112.3.678. PMID 9676983
- [Background] Johnson AW. Characterizing ingestive behavior through licking microstructure: Underlying neurobiology and its use in the study of obesity in animal models. Int J Dev Neurosci. 2018 Feb;64:38-47. doi: 10.1016/j.ijdevneu.2017.06.012. Epub 2017 Jul 3. PMID 28684308
- [Derived] Gero D, File B, Alceste D, Frick LD, Serra M, Ismaeil AE, Steinert RE, Spector AC, Bueter M. Microstructural changes in human ingestive behavior after Roux-en-Y gastric bypass during liquid meals. JCI Insight. 2021 Aug 9;6(15):e136842. doi: 10.1172/jci.insight.136842. PMID 34369388